CLINICAL TRIAL: NCT02881996
Title: Impact of IV Acetaminophen on Post-operative Pain After Laparoscopic Appendectomy for Perforated Appendicitis: A Prospective Randomized Trial
Brief Title: The Impact of IV Acetaminophen on Pain After Appendectomy for Perforated Appendicitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Mercy Hospital Kansas City (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 13100328
Record Dates: First submitted 2016-01-18; First posted 2016-08-29 (Estimated); Results first posted 2021-01-12 (Actual); Last update posted 2021-01-12 (Actual); Status verified 2020-12

CONDITIONS: Perforated Appendicitis
Keywords: appendicitis; pain; perforation
MeSH Terms: conditions — Appendicitis; Pain | interventions — Acetaminophen; Ketorolac; Ketorolac Tromethamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- IV tylenol (Experimental): Post-operatively, all patients will be placed on a standard patient/nurse controlled analgesia (PCA) according to our pain service protocol which included ketorolac. A 3 hours after first dose of ketorolac, patients in the acetaminophen arm will then receive scheduled 10mg/kg of IV acetaminophen every 6hrs for a total of 3 days in between doses of ketorolac. PCA Pumps will be discontinued with the return of bowel function and transition to oral intake in all patients as per the current protocol. If a patient in the acetaminophen arm is transitioned off of PCA prior to 3 days, IV acetaminophen will be stopped at that time as well. Patients in the control group only may receive oral/rectal acetaminophen as needed for treatment of fevers.
  Interventions: Drug: IV tylenol; Drug: Ketorolac
- No IV tylenol (Active Comparator): Same as above without IV tylenol.
  Interventions: Drug: No IV tylenol; Drug: Ketorolac

INTERVENTIONS:
Drug: IV tylenol — IV tylenol given scheduled in addition to standard PCA
  Other Names: acetaminophen,
  Arms: IV tylenol
Drug: No IV tylenol — No additional IV Tylenol given
  Arms: No IV tylenol
Drug: Ketorolac — both groups receive as part of our standard postop pain protocol after all operations
  Other Names: toradol

SUMMARY:
The objective of this study is to evaluate two standard post-operative pain regimens routinely used after laparoscopic appendectomy for perforated appendicitis. The investigators hypothesize that the use of intravenous (IV) acetaminophen in addition to IV ketorolac with narcotic pain pump will decrease time to transition off patient/nurse controlled analgesia (PCA) to oral pain medications.

DETAILED DESCRIPTION:
To assess pain control, patient and family perception of pain control, time to return of bowel function defined as passage of first flatus (in days), doses of anti-emetic medications, doses of narcotic pain medications, time to toleration of regular diet (in days), narcotic associated adverse effects (nausea, emesis, respiratory depression, constipation), length of stay, and overall hospital cost in admission.

Post-hospitalization the investigators will assess complications including number and reasons for emergency visits and abscess formation, length of post-hospitalization analgesic use, length of post-hospitalization narcotic use, and time to return to school.

ELIGIBILITY:
Inclusion Criteria:

* All patients ages 2-17 years old undergoing laparoscopic appendectomy at CMH found to have perforated appendicitis.

Exclusion Criteria:

* Non-perforated appendicitis
* Normal appendix at the time of operation or other associated conditions causing abdominal pain
* Patients with history of chronic pain
* Known underlying liver disorders
* Known allergy to pain medication in protocol
* Non-English speaking

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 90 (Actual)
Dates: Start 2014-06; Primary Completion 2016-06 (Actual); Study Completion 2016-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shawn D St. Peter, MD, Principal Investigator — Children's Mercy Hospital Kansas City
Locations (1):
- Children's Mercy Hospital, Kansas City, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | IV Tylenol | No IV Tylenol
Started | 45 | 45
Completed | 39 | 43
Not Completed | 6 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | IV Tylenol | No IV Tylenol | Total
Number analyzed (Participants) | 39 | 43 | 82
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 39 | 43 | 82
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 10.9 [6.9 to 14.9] | 9.6 [5.6 to 13.6] | 10.25 [5.6 to 14.9]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 13 | 27
  Male | 25 | 30 | 55
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 39 | 43 | 82

OUTCOME MEASURES:

1. Primary Outcome: Time Until PCA Discontinued After the Operation
Description: The investigators hypothesize that the use of intravenous (IV) acetaminophen in addition to IV ketorolac with narcotic pain pump will decrease time to transition off PCA/NCA to oral pain medications.
Time Frame: 4 days
Measure: Mean (95% Confidence Interval); unit: hours
Arm/Group | IV Tylenol | No IV Tylenol
Number analyzed (Participants) | 39 | 43
hours | 76.4 [43.9 to 108.9] | 86.7 [37.4 to 136]

2. Secondary Outcome: Postoperative Duration of Hospital Stay
Description: The investigators will measure postoperative time to discharge
Time Frame: 1 week
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | IV Tylenol | No IV Tylenol
Number analyzed (Participants) | 39 | 43
days | 3.9 [3.1 to 5.9] | 4.5 [3.1 to 6.1]

ADVERSE EVENTS:
Time Frame: Duration of length of stay up to one week.
Arm/Group | IV Tylenol | No IV Tylenol
All-Cause Mortality (participants affected / at risk) | 0/39 | 0/43
Serious Adverse Events (participants affected / at risk) | 0/39 | 0/43
Other Adverse Events (participants affected / at risk) | 0/39 | 0/43

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No